CLINICAL TRIAL: NCT02650505
Title: A Randomized, Controlled Study to Evaluate the Sensitizing Potential of LEO 43204 Gel and Gel Vehicle in Healthy Volunteers Using a Repeat Insult Patch Test Design
Brief Title: A Clinical Study to Evaluate the Sensitizing Potential of LEO 43204 Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LP0084-1230
Record Dates: First submitted 2015-12-04; First posted 2016-01-08 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2017-07

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — LEO 43204

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 43204 (Experimental): LEO 43204 will be applied topically to the skin under open conditions 10 times
  Interventions: Drug: LEO 43204
- LEO 43204 vehicle (Placebo Comparator): LEO 43204 vehicle will be applied topically to the skin under open conditions 10 times
  Interventions: Drug: LEO 43204 Vehicle

INTERVENTIONS:
Drug: LEO 43204
  Arms: LEO 43204
Drug: LEO 43204 Vehicle
  Arms: LEO 43204 vehicle

SUMMARY:
This is a randomized, single-center, controlled, within-subject comparison study assessing the sensitization potential of the investigational product, LEO 43204 gel under open conditions in healthy volunteers.

LEO 43204 Gel and Vehicle Gel will be applied to adjacent sites on the infrascapular area of the back. Evaluation of dermal reactions at the application sites will be assessed clinically using a visual scale that rates the degree of erythema, edema and other signs of cutaneous irritation.

Following induction, subjects will have a 10 to 14-day Rest Phase, after which they will enter the Challenge Phase, which consists of one 48-hour application to a naive site on the opposite side of the back. Observations at the naive site during Challenge and the patterns of reactivity during the Induction Phase will provide a basis for an interpretation of contact sensitization.

A total of 10 applications will be made over a period of approximately 6-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events;
2. Fitzpatrick skin types I-IV (due to lack of safety data for the investigational product in darker skin types);
3. Complete a Medical Screening form as well as a Medical Personal History form;

Exclusion Criteria:

1. Have any visible skin disease at the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction;
2. Are not willing to refrain from using topical/systemic analgesics for 72 hours prior to and during the study (daily use of 81 mg aspirin is acceptable and occasional use of acetaminophen will be permitted);
3. Are using systemic/topical corticosteroids for 3 weeks prior to and during the study, or systemic/topical antihistamines for 72 hours prior to and during the study;
4. Are using medication which, in the opinion of the investigative personnel, will interfere with the study results, including anti-inflammatory medications;
5. Are unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions, or similar products on the back during the study;
6. Have psoriasis and/or active atopic dermatitis/eczema;
7. Have damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The determination of dermal sensitization will be based on LSRs and confirmed at a Rechallenge. If recurrence in Rechallenge is equivalent to or more severe than observed at challenge it will be considered indicative of a sensitization reaction. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research Inc., Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en